CLINICAL TRIAL: NCT02647567
Title: Can Caffeine Intake Combined With Aerobic Exercise Leads to Cognitive Improvement and Psychomotor Performance in Trained Individuals?
Brief Title: Caffeine Intake and Additive Effects on Cognition
Acronym: Caffeine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Alberto Souza de Sá Filho, Doctorade in Mental Health, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: UNIVERSO-03
Record Dates: First submitted 2015-12-05; First posted 2016-01-06 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2016-01

CONDITIONS: Healthy
Keywords: Cognitive; Aerobic Exercise; Performance
MeSH Terms: interventions — Caffeine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Caffeine Intake (Experimental): The experimental group ingest 500 mg of caffeine before (60 min) aerobic exercise (procedure double blind), and perform a battery of neuropsychological and psychomotor tests. 1 min and 30 min after the exercise the subjects perform a new battery of neuropsychological and psychomotor tests.
  Interventions: Other: Caffeine Intake
- Placebo Intake (Placebo Comparator): The control group ingest 500 mg of placebo before (60 min) aerobic exercise (procedure double blind), and perform a battery of neuropsychological and psychomotor tests. 1 min and 30 min after the exercise the subjects perform a new battery of neuropsychological and psychomotor tests.
  Interventions: Other: Placebo Intake

INTERVENTIONS:
Other: Caffeine Intake — The experimental group ingest 500 mg of caffeine before (60 min) aerobic exercise (procedure double blind), and perform a battery of neuropsychological and psychomotor tests. 1 min and 30 min after the exercise the subjects perform a new battery of neuropsychological and psychomotor tests.
  Other Names: Caffeine
  Arms: Caffeine Intake
Other: Placebo Intake — The control group ingest 500 mg of placebo before (60 min) aerobic exercise (procedure double blind), and perform a battery of neuropsychological and psychomotor tests. 1 min and 30 min after the exercise the subjects perform a new battery of neuropsychological and psychomotor tests.
  Other Names: Placebo
  Arms: Placebo Intake

SUMMARY:
Caffeine is a methylxanthine commonly consumed by the population for their psychostimulant properties, and their intake when in moderate doses seem to produce positive effects on stress, mood and memory. So, understanding that a positive effect of aerobic exercise can be displayed also on cognition, as caffeine, when in proper proportions, the investigators do not know if the joining of the two strategies into a single activity would be able to promote additional effects enhancing cognitive processes related to memory, attention, and motor reaction time.

DETAILED DESCRIPTION:
Determine if 500 mg of caffeine can generate additional effects to 30 minutes of aerobic exercise enhancing cognitive memory tasks (Rey Auditory Verbal Learning Test - RAVLT), attention (sustained attention span; working speed; Percentual of errors by confusion) and simple reaction time (SRT).

ELIGIBILITY:
Inclusion Criteria:

* Fighting men
* Low levels of consumption of caffeine daily

Exclusion Criteria:

* Use more than 400 mg caffeine day
* Mental diseases
* Cognitive deficits

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-05; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Simple Reaction Time | Acute Change from Baseline Psychomotor test to 1 min after aerobic exercise, and after 30 min
Rey Auditory Verbal Learning Test | Acute Change from Baseline Cognitive test to 1 min after aerobic exercise, and after 30 min
Sustained Attention Test | Acute Change from Baseline Cognitive test to 1 min after aerobic exercise, and after 30 min

CONTACTS AND LOCATIONS:
Overall Officials: Sérgio Machado, PhD, Study Director — Salgado de Oliveira University

IPD SHARING:
Plan to Share IPD: Undecided